CLINICAL TRIAL: NCT04776577
Title: Assessment of Coronary Pressure Using the Combined Guidewire and Catheter Wirecath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Cavis Technologies AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0100P
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2021-02

CONDITIONS: Coronary Disease
Keywords: coronary disease; fractional flow reserve; coronary flow reserve; pressure wire
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: Results from simultaneous measurements with two wires will be graphically showed using the Bland-Altman plot and reported in terms of intraclass correlation coefficient (ICC). Also, whether a theoretical correction for the expected hydrostatic pressure error (0.77 mmHg per cm height difference) at the distal pressure measurement site (Pd) accounts for the difference in FFR during simultaneous measurements will be explored, and a corrected ICC reported. A two-sided p-value of <0.05 will be considered to be significant, when applicable.
  The Pearson's correlation coefficient will be also calculated considering the Wirecath FFR value in comparison to the FFR value made with the regular wire with and without correction for hydrostatic error.
  For the CFR values, the Pearson's correlation coefficient will be used to determine the relation between the bolus-thermo CFR, absolute-flow CFR, Echo CFR and the pressure-derived CFR in the LAD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Other): Group 1 and group 2 will be recruited and assessed in parallel at the discretion of the treating physician, based on the characteristics of the patient. Group 3 will be recruited from suitable patients in group 1 and 2.
  Simultaneous measurements study (group 1) Regular study group (group 2) Echocardiography-CFR group (group 3)
  Interventions: Device: Wirecath@ and Abbott PressureWire® (20 patients); Device: Wirecath® (20 patients); Device: Coronary flow reserve

INTERVENTIONS:
Device: Wirecath@ and Abbott PressureWire® (20 patients) — Simultaneous FFR measurements with Wirecath@ and Abbott PressureWire®
Device: Wirecath® (20 patients) — FFR measurement with Wirecath® only
Device: Coronary flow reserve — Pressure derived CFR with Wirecath®, Thermodilution CFR with Abbott PressureWire®, Absolut flow CFR with Abbott PressureWire® and Hexacath Rayflow catheter®, Non-invasive echo derived CFR

SUMMARY:
In summary, the purpose of the study is to evaluate whether the Wirecath device can be used as a standard pressure wire in a safe and efficient way.

DETAILED DESCRIPTION:
Simultaneous measurements study (group 1) This group will be recruited and assessed in parallel with recruitment to group 2 at the discretion of the treating physician, based on the resource availability in the cath lab.

In the simultaneous measurements study group, measurements will be collected from a Wirecath® and a regular sensor-tipped pressure wire in the same position in the coronary artery at the same time (simultaneously). The regular wire to be used is the market leading Abbott PressureWire®.

By comparing the pressure measurements (Pd) from Wirecath® and from a regular sensor-tipped wire, we intend to examine if the pressure reported by the two wires deviate in any way. If a deviation exists, the hydrostatic error, caused by the height difference between the positions of Pa and Pd when using a sensor-tipped wire, will be assessed.

In FFR-negative patients, after removal of the Wirecath®, the Abbott PressureWire® is used in LAD

* first to measure CFR by saline bolus injections and thermodilution during rest and hyperemia (Bolus-thermo CFR) and
* second together with a Hexacath/Rayflow@ infusion catheter and a saline infusion pump to measure absolute flow during rest and hyperemia that will be used to calculate CFR (Absolute-flow CFR).

Wirecath will be used for PCI when indicated and performance documented by follow-up questions to the users.

Regular study group (group 2) In the regular use study group, the Wirecath® is to be used as a regular pressure measurement tool, replacing the regularly used pressure wire.

Pressure measurement results will be collected.

Wirecath® will be used for PCI when indicated and performance documented by follow-up questions to the users.

In FFR-negative patients, after removal of the Wirecath®, the Abbott PressureWire® is used in LAD

* first to measure CFR by saline bolus injections and thermodilution during rest and hyperemia (Bolus-thermo CFR) and
* second together with a Hexacath/Rayflow® infusion catheter and a saline infusion pump to measure absolute flow during rest and hyperemia that will be used to calculate CFR (Absolute-flow CFR).

Echocardiography-CFR group (group 3) Patients from group 1 and group 2 that have undergone Bolus-thermo and Absolute-flow CFR measurements, will be recruited to group 3. In this group echocardiography-CFR (Echo CFR) will be measured within 14 days. The echocardiography is performed according to the standard procedure of the hospital. The correlation between the methods will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18yrs age)
* Informed consent given
* Patients with result from diagnostic angiography
* Indication for coronary pressure assessment

Exclusion Criteria:

* Patients with known Heparin-Induced Thrombocytopenia (HIT) or allergy to heparin.
* Inability to tolerate Adenosine
* Any condition, e.g. unstable health, which in the opinion of the investigator makes the patient unsuitable for inclusion (Decision documented in inclusion log).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Safety of the Wirecath® will be assessed through the frequency and severity of all adverse events | 30-60 minutes
  The safety of the Wirecath@ will be assessed through the frequency and severity of all adverse events reported for study subjects after the completion of the pressure measurement and PCI. The primary endpoint will be achieved when the device has been used on enrolled patients and required measurements have been taken.

SECONDARY OUTCOMES:
Comparison with Abbott pressure wire | 30-60 minutes
  comparing the Wirecath measurement values with the measurement values of a regular sensor-tipped pressure guidewire during simultaneous measurements in the same vessel.
Comparing pressure-derived coronary flow reserve (CFR) with bolus-thermo CFR, absolute flow CFR and non-invasive doppler derived CFR | 14 days
  In FFR negative LADs, comparing the Wirecath® pressure-derived CFR values with CFR derived from thermodilution, absolute flow and echocardiography-CFR values. This secondary endpoint will be achieved if these values correlate

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Angerås, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Ramunddal T, Dworeck C, Torild P, Andreen S, Gan LM, Hirlekar G, Ioanes D, Myredal A, Odenstedt J, Petursson P, Pylova T, Topel F, Volz S, Hilmersson M, Redfors B, Angeras O. Safety and Feasibility Using a Fluid-Filled Wire to Avoid Hydrostatic Errors in Physiological Intracoronary Measurements. Cardiol Res Pract. 2024 Jan 2;2024:6664482. doi: 10.1155/2024/6664482. eCollection 2024. PMID 38204600